CLINICAL TRIAL: NCT03852056
Title: The Clinical Investigation of a New Toothpaste Containing SnF as Compared to Colgate Fluoride Toothpaste in Reducing Plaque and Gingivitis - a Six-month Study in China
Brief Title: The Clinical Investigation of a New Toothpaste Containing Stannous Fluoride as Compared to a Commercially Available Fluoride Toothpaste in Reducing Plaque and Gingivitis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Colgate Palmolive (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CRO-2017-02-GIN-SNDZ-YPZ
Record Dates: First submitted 2019-02-21; First posted 2019-02-22 (Actual); Last update posted 2019-02-22 (Actual); Status verified 2019-01

CONDITIONS: Dental Plaque; Gingivitis
MeSH Terms: conditions — Dental Plaque; Gingivitis

STUDY DESIGN:
Intervention Model Description: Tooth brushing study. Subjects brush their whole mouth 2x/day for 1 minute each time. The study duration is 6 months
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: All clinical product will be in a plain white toothpaste tube or over wrapped with white laminate material to conceal any product identity. All study treatments will have a clinical label attached that contains study information and a unique product code.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MFP Fluoride toothpaste (Placebo Comparator): Commercially available, monofluorophosphate (MFP) toothpaste. Fluoride level is 0.76%
  Interventions: Drug: MFP Fluoride toothpaste
- Stannous Fluoride Toothpaste (Experimental): New toothpaste containing 0.454% stannous fluoride.
  Interventions: Drug: Stannous fluoride toothpaste

INTERVENTIONS:
Drug: MFP Fluoride toothpaste — Whole mouth brushing with a toothpaste, 2 times/day for 1 minute each time for the duration of the study,
  Other Names: Colgate Great Regular Flavor toothpaste
  Arms: MFP Fluoride toothpaste
Drug: Stannous fluoride toothpaste — Whole mouth brushing with a toothpaste, 2 times/day for 1 minute each time for the duration of the study,
  Arms: Stannous Fluoride Toothpaste

SUMMARY:
The objective of this study is to evaluate the clinical efficacy of a new toothpaste containing stannous fluoride (SnF) as compared to Colgate Fluoride Toothpaste in reducing gingivitis and dental plaque.

DETAILED DESCRIPTION:
This is a 6 month, take home, tooth brushing research study to evaluate a new toothpaste.

Qualified subjects will be enrolled and randomized to either one of the two study groups based on their initial Plaque and Gingivitis scores. Subjects will be instructed to use the products according to the instructions provided. Subjects will return to the dental office for evaluation after three and six months of product use. All subjects will be followed for adverse events throughout the study.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects, ages 18-70, inclusive.
2. Availability for the six-month duration of the clinical research study.
3. Good general health.
4. Minimum of 20 uncrowned permanent natural teeth (excluding third molars).
5. Initial gingivitis index of at least 1.0 as determined by the use of the Loe and Silness Gingival Index.
6. Initial plaque index of at least 1.5 as determined by the use of the Quigley and Hein Plaque Index (Turesky Modification).
7. Signed Informed Consent Form.

Exclusion Criteria:

1. Presence of orthodontic bands.
2. Presence of partial removable dentures.
3. Tumor(s) of the soft or hard tissues of the oral cavity.
4. Advanced periodontal disease (purulent exudate, tooth mobility, and/or extensive loss of periodontal attachment or alveolar bone).
5. Five or more carious lesions requiring immediate restorative treatment.
6. Antibiotic use any time during the one-month period prior to entry into the study.
7. Participation in any other clinical study or test panel within the one month prior to entry into the study.
8. Dental prophylaxis during the past two weeks prior to baseline examinations.
9. History of allergies to oral care/personal care consumer products or their ingredients.
10. On any prescription medicines that might interfere with the study outcome.
11. An existing medical condition that prohibits eating or drinking for periods up to 4 hours.
12. History of alcohol or drug abuse.
13. Self-reported pregnant or lactating subjects.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 98 (Actual)
Dates: Start 2017-05-25 (Actual); Primary Completion 2017-12-07 (Actual); Study Completion 2017-12-07 (Actual)

PRIMARY OUTCOMES:
Dental Plaque Scores | Baseline
  Quigley-Hein, Turesky Modification Index. Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Dental Plaque Scores | 3 month
  Quigley-Hein, Turesky Modification Index. Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Dental Plaque Scores | 6 month
  Quigley-Hein, Turesky Modification Index. Units on a scale 0 to 5 (0 = no plaque, 1 = separate flecks of plaque on the tooth, 2 = a thin continuous band of plaque, 3 = a band of plaque up to one-third of the tooth, 4 = plaque covering up to two thirds of the of the tooth, 5 = plaque covering two-thirds or more of the crown of the tooth)
Gingivitis Scores | Baseline
  Loe & Silness Gingival Index. Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Gingivitis Scores | 3 months
  Loe & Silness Gingival Index. Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)
Gingivitis Scores | 6 months
  Loe & Silness Gingival Index. Units on a scale 0 to 3 (0 = no inflammation, 1 = Mild inflammation-slight change in color and little change in texture 2 = Moderate inflammation-moderate glazing, redness, edema and hypertrophy. Tendency to bleed upon probing. 3 = Severe inflammation-marked redness and hypertrophy. Tendency to spontaneous bleeding)

CONTACTS AND LOCATIONS:
Locations (1):
- West China Dental Institute of Chengdu, Chengdu, Sichuan, China

IPD SHARING:
Plan to Share IPD: No